CLINICAL TRIAL: NCT00750906
Title: The Muscle Biochemical, Serum Potassium and Cardiovascular Changes After Succinylcholine in Patients Undergoing Electroconvulsive Therapy.
Brief Title: ECT/Succinylcholine: Biochemical, Serum and Cardiovascular Changes
Status: Terminated | Type: Observational
Why Stopped: Study on hold since 2009. Awaiting FDA approval of Sugammdex to complete second arm of study.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H898-32701
Record Dates: First submitted 2008-09-09; First posted 2008-09-11 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will be conducted to determine the pharmacodynamics, cardiovascular and biochemical effects of succinylcholine when given during electroconvulsive therapy. (ECT). This is a single center, prospective, study in patients who will be receiving ECT as indicated and prescribed by their psychiatrist. The study will be performed twice on each patient, 48-72 hours apart during consecutively scheduled ECT procedures.

DETAILED DESCRIPTION:
Patients will receive the anesthetic that is traditionally given which includes appropriate doses of succinylcholine. Serum potassium and creatinine phosphokinase (CK) levels will be determined pre and post anesthesia; serum and urine myoglobin will be determined post anesthesia. Vital signs data [i.e., heart rate (arrhythmias) and arterial blood pressure] will be compared pre and post anesthesia. In addition patients will be asked about the presence of muscle pain (myalgia) 1 hour before discharge from the recovery room and the following day post ECT.

ELIGIBILITY:
Inclusion Criteria:

1. A male or non-pregnant female aged 18 years and older
2. American Society of Anesthesiologists physical status 1, 2, 3
3. Scheduled to undergo electroconvulsive therapy under general anesthesia
4. Have given written informed consent

Exclusion Criteria:

1. Pregnant or nursing
2. Any patient in the study investigators opinion who may not be suitable for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing electroconvulsive therapy.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2008-10; Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Miller, MD, Study Director — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States